CLINICAL TRIAL: NCT06254859
Title: Intraoperative Neuromuscular Monitoring and Its Impact on Pre- and Postoperative Acoustic Outcomes in Thyroid Surgery
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Director, Head of Thyroid Surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Other Study IDs: THYRO-SOUND2024
Record Dates: First submitted 2024-01-30; First posted 2024-02-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Thyroid Cancer; Thyroid Cancer, Papillary
Keywords: acoustic analysis; thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Normal Signal Group.: During the surgical procedure, there was no occurrence of a decrease in recurrent laryngeal nerve signals or a decrease of less than 10%.
  Interventions: Procedure: Traditional thyroid surgery.
- Signal Decrease 10-50%.: During the surgical procedure, the signal of the recurrent laryngeal nerve decreased by 10-50%.
  Interventions: Procedure: Traditional thyroid surgery.
- Signal Decrease 50-90%.: During the surgical procedure, the signal of the recurrent laryngeal nerve decreased by 50-90%.
  Interventions: Procedure: Traditional thyroid surgery.
- Signal Absence Group.: During the surgical procedure, the signal of the recurrent laryngeal nerve decreased by more than 90% or completely disappeared.
  Interventions: Procedure: Traditional thyroid surgery.

INTERVENTIONS:
Procedure: Traditional thyroid surgery. — The patient undergoes traditional thyroid surgery with concurrent intraoperative nerve monitoring technology.

SUMMARY:
This study examines the impact of intraoperative recurrent laryngeal nerve monitoring signal changes on the postoperative voice quality of thyroid surgery patients. By analyzing extensive surgical data and postoperative voice recordings, the investigation seeks to identify patterns in the variations of these signals and their correlation with voice quality outcomes. The goal is to enhance clinical understanding and surgical practices, allowing for more precise assessments of nerve function, informed surgical interventions, and improved postoperative patient well-being.

DETAILED DESCRIPTION:
This research project conducts a detailed exploration into the fluctuations of intraoperative recurrent laryngeal nerve monitoring signals during thyroid surgery and their subsequent effects on the voice quality of patients after surgery. The study meticulously analyzes a comprehensive dataset comprised of surgical records and voice analyses conducted before and after the procedure. The primary objective is to pinpoint specific trends and changes in the nerve monitoring signals and to determine how these alterations correlate with the postoperative acoustic characteristics of patients' voices. By establishing a clear link between intraoperative signal dynamics and postoperative voice outcomes, the investigation aims to advance the field of thyroid surgery. This includes providing surgeons with critical insights for the precise evaluation of recurrent laryngeal nerve functionality, enabling targeted interventions during operations, and ultimately contributing to the enhancement of patients' quality of life following surgery. Through this rigorous analysis, the study seeks to contribute valuable knowledge to the surgical community, facilitating improved patient care and outcomes in thyroid surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years old.
* Planned conventional unilateral thyroid lobectomy + isthmus resection + central compartment lymph node dissection.

Exclusion Criteria:

* History of past head and neck surgeries.
* Pronunciation system defect and disorder history.
* History of vocal cord polyps or nodules.
* History of upper respiratory tract infection in the 2 weeks before surgery or postoperative infection history.
* History of neurological disorders.
* Abnormalities in the throat.
* Preoperative damage to throat morphology or motor function.
* Preoperative functional voice or language disorders, noticeable hoarseness, or difficulty in pronunciation.
* Pre- and postoperative laryngoscopic examination showing vocal cord paralysis and arytenoid joint dislocation.
* Neurological disorders causing abnormal throat function.
* Patient unable to cooperate with VHI (Voice Handicap Index) assessment and voice spectrum examination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with thyroid cancer who are planned to undergo traditional surgical treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative electromyographic signals. | During the surgery, record R1 and V1 signals when initially identifying the recurrent laryngeal nerve or vagus nerve. After the surgery, record R2 and V2 signals upon re-identification of the recurrent laryngeal nerve or vagus nerve.
  Recording intraoperative electromyographic signals, including vagus nerve V1 and V2 signals, recurrent laryngeal nerve R1 and R2 signals.
Voice analysis data(SPL) | Before the surgery, 2 weeks after the surgery, 2 months after the surgery, 4 months after the surgery, and 6 months after the surgery.
  Recording data(SPL) of voice tests before and after the surgery, sound pressure level in dB(A)
Voice analysis data(F0) | Before the surgery, 2 weeks after the surgery, 2 months after the surgery, 4 months after the surgery, and 6 months after the surgery.
  Recording data(F0) of voice tests before and after the surgery, F0 in Hz
Voice analysis data(Jitter) | Before the surgery, 2 weeks after the surgery, 2 months after the surgery, 4 months after the surgery, and 6 months after the surgery.
  Recording data(Jitter) of voice tests before and after the surgery, Jitter in percentage
Voice analysis data(Shimmer) | Before the surgery, 2 weeks after the surgery, 2 months after the surgery, 4 months after the surgery, and 6 months after the surgery.
  Recording data(Shimmer) of voice tests before and after the surgery, Shimmer in percentage

SECONDARY OUTCOMES:
RBH | Before the surgery, 2 weeks after the surgery, 2 months after the surgery, 4 months after the surgery, and 6 months after the surgery.
  Conducted by an otolaryngologist, the RBH assessment includes R (Roughness), B (Breathiness), and H (Hoarseness).
VHI-30 | Before the surgery, 2 weeks after the surgery, 2 months after the surgery, 4 months after the surgery, and 6 months after the surgery.
  Voice Handicap Index, including a scale with 30 items.The full, non-abbreviated title of the VHI-30 scale is the "Voice Handicap Index-30," and it is translated as the "Voice Disorder Severity Index." The scale ranges from a minimum score of 0 to a maximum of 120, with higher scores indicating poorer outcomes.
Neural Width | During surgery.
  Recorded width of the recurrent laryngeal nerve in millimeters.
Is there branching | During surgery.
  Note if the recurrent laryngeal nerve branches.
Number of neural branches | During surgery.
  If there are branches in the recurrent laryngeal nerve, record the number of branches.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No